CLINICAL TRIAL: NCT01367990
Title: Alopecia Prevention Trial of Topical Vasoconstrictor Therapy in Head and Neck Cancer Patients Treated With Intensity Modulated Radiotherapy (IMRT)
Brief Title: Exploratory Study of Norepinephrine to Prevent Alopecia in Head and Neck Cancer Patients Treated With Radiotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study site has terminated the study due to the complexity of the study
Sponsor: ProCertus BioPharm, Inc (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PC-5
Record Dates: First submitted 2011-06-05; First posted 2011-06-07 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Alopecia; Radiodermatitis
Keywords: alopecia; hair loss; prevention; radiotherapy; head & neck cancer; radiodermatitis; radiation dermatitis; radiation-induced alopecia
MeSH Terms: conditions — Alopecia; Radiodermatitis; Head and Neck Neoplasms | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norepinephrine (Experimental)
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — The occipital scalp zone at risk for alopecia will be identified. The norepinephrine treatment site will be randomized to receive consistent treatment of one half of the scalp "risk zone." Approximately 1.6 mL of a 400 mM norepinephrine solution will be applied topically to the norepinephrine site approximately 20 minutes prior to each radiation treatment, and placebo will be applied to the contralateral side (30-35 treatments).
  Other Names: Noradrenaline

SUMMARY:
The study will evaluate the safety of topical norepinephrine in head and neck cancer patients who are receiving treatment with intensity modulated radiotherapy (IMRT).

The study will also provide information about whether topical norepinephrine can prevent or decrease the severity of the radiation-induced alopecia experienced by these patients.

ELIGIBILITY:
Inclusion Criteria:

* be ≥ 18 years of age with documented pathological diagnosis of H&N (head and neck) cancer.
* planned to receive H&N region IMRT treatment in which the mean dose to the dermis in the scalp risk zone (isodose plan) is estimated to be at least 20 Gy.
* have a palpable nuchal prominence (external occipital protuberance)
* have the ability to understand the informed consent document.
* be able to comply with protocol schedule.
* have a negative serum pregnancy test if a female of childbearing potential.
* consent to utilize medically acceptable methods of contraception throughout the study if of childbearing potential.
* be treated with IMRT alone or with concurrent platinum based chemotherapy
* receive definitive treatment for oropharyngeal squamous cell carcinoma

Exclusion Criteria:

* with clinical or radiographic evidence of adenopathy to the high level V posterior cervical nodes, post-auricular or occipital cervical nodal stations
* planned to receive H&N region treatment in which the mean dose to the dermis in the scalp risk zone (isodose plan) is estimated to exceed 50Gy
* with underlying active untreated cardiac disease (e.g. arrhythmia)
* receiving concurrent chemotherapy other than single agent platinum based
* with generalized skin disorders that have required treatment within the past 6 months.
* with connective tissue disorders
* with unhealed wounds or scars in the study area
* with rashes, ulcerations, or poorly healed scars in the treatment area
* with a known allergy to norepinephrine
* with a known clinically significant abnormal ECG (electrocardiogram) within the past 6 months.
* taking MAO (monoamine oxidase) inhibitors or antidepressants of the triptyline or imipramine types
* taking β-blockers
* with NCI-CTCAE Version 4.0 grade 2 or higher hypertension at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Safety of daily topical application of norepinephrine to the radiation field. | Safety will be assessed during the study (6-7 weeks) and at follow-up visits approximately 2 and 4 weeks after the end of the treatment period.
  The primary safety hypothesis is that there will be that there will be little or no scalp irritation associated with the application of the topical norepinephrine and that there will be no systemic effects secondary to transdermal absorption.

SECONDARY OUTCOMES:
Efficacy of daily topical application of norepinephrine to the radiation field. | Efficacy will be assessed during the study (6-7 weeks) and at follow-up visits approximately 2 and 4 weeks after the end of the treatment period
  The primary efficacy hypothesis is that areas of the scalp that are treated with topical norepinephrine immediately prior to intensity modulated radiotherapy (IMRT) will have less severe alopecia than scalp sites that are not treated with topical norepinephrine and that receive only placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Rao, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States